CLINICAL TRIAL: NCT03244839
Title: Prevalence of Major Nutrients Deficiency in Diabetic Patient Before and After Bariatric Surgery
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Min-Sheng General Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2016007
Record Dates: First submitted 2017-07-28; First posted 2017-08-10 (Actual); Last update posted 2017-08-10 (Actual); Status verified 2017-07

CONDITIONS: Diabetic Patient Before and After Bariatric Surgery; Nutrition Deficiency(VitB1 VitB12.Ca.Fe)
MeSH Terms: interventions — Bariatric Surgery

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: bariatric surgery — bariatric surgery

SUMMARY:
The increasing demand of bariatric surgery requires ongoing improvement of the preoperative and post-operative care of morbidly obese patients. Outcome reporting in bariatric surgery mainly focuses on weight loss, improvement of co-morbidities and quality of life. Post-operative nutritional deficiencies are a complication of bariatric surgery, in particular after malabsorptive procedures. Deficiencies of protein, iron and vitamins B12 and D are frequently reported and may occur despite supplementation. Morbid obesity itself is associated with nutritional deficiencies as well, which become worsening after bariatric surgery. The occurrence of nutritional deficiencies has been reported in the literature but not in Taiwan. The goal of the current study is to determine the prevalence and incidence of nutritional deficiencies in diabetic patients underwent bariatric surgery and receiving standard supplementation in Taiwan.

DETAILED DESCRIPTION:
The increasing demand of bariatric surgery requires ongoing improvement of the preoperative and post-operative care of morbidly obese patients. Outcome reporting in bariatric surgery mainly focuses on weight loss, improvement of co-morbidities and quality of life. Post-operative nutritional deficiencies are a complication of bariatric surgery, in particular after malabsorptive procedures. Deficiencies of protein, iron and vitamins B12 and D are frequently reported and may occur despite supplementation. Morbid obesity itself is associated with nutritional deficiencies as well, which become worsening after bariatric surgery. The occurrence of nutritional deficiencies has been reported in the literature but not in Taiwan. The goal of the current study is to determine the prevalence and incidence of nutritional deficiencies in diabetic patients underwent bariatric surgery and receiving standard supplementation in Taiwan

ELIGIBILITY:
Inclusion Criteria:

* Age: 20~65
* Diabetic patients underwent bariatric surgery in MSGH

Exclusion Criteria:

* Pregnancy
* Cancer on treatment
* Uncontrolled psychiatric disease
* Drug or alcohol abuser

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Diabetic patients underwent bariatric surgery in MSGH
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2016-01; Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Prevalence of major nutrients deficiency in diabetic patient before and after bariatric surgery | 3 years
  Prevalence of major nutrients deficiency in diabetic patient before and after bariatric surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Min sheng general hospital, Taoyuan, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Shiffman ML, Sugerman HJ, Kellum JM, Moore EW. Changes in gallbladder bile composition following gallstone formation and weight reduction. Gastroenterology. 1992 Jul;103(1):214-21. doi: 10.1016/0016-5085(92)91115-k. PMID 1612328
- [Result] Shiffman ML, Sugerman HJ, Kellum JM, Brewer WH, Moore EW. Gallstone formation after rapid weight loss: a prospective study in patients undergoing gastric bypass surgery for treatment of morbid obesity. Am J Gastroenterol. 1991 Aug;86(8):1000-5. PMID 1858735
- [Result] Williams C, Gowan R, Perey BJ. A Double-Blind Placebo-controlled Trial of Ursodeoxycholic Acid in the Prevention of Gallstones during Weight Loss after Vertical Banded Gastroplasty. Obes Surg. 1993 Aug;3(3):257-259. doi: 10.1381/096089293765559278. PMID 10757929